CLINICAL TRIAL: NCT03987529
Title: Comparison of Effects of Volatile and Intravenous Anesthetics on Pupillary Function During General Anesthesia in Children; a Prospective Observational Study.
Brief Title: Effects of Volatile and Intravenous Anesthetics on Pupillary Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, professor, Seoul National University Hospital
Other Study IDs: H1906-096-1040
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Pupillary Functions, Abnormal
MeSH Terms: conditions — Pupil Disorders | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sevoflurane+Remifentanil: Using inhalent agent(Sevoflurane), continuous infusion of Remifentanil
  Interventions: Other: sevoflurane
- Propofol+Remifentanil: Using continuous infusion of Propofol and Remifentanil
  Interventions: Other: propofol

INTERVENTIONS:
Other: sevoflurane — volatile anesthetic
  Groups: Sevoflurane+Remifentanil
Other: propofol — intravenous anesthetic
  Groups: Propofol+Remifentanil

SUMMARY:
To compare of effects of volatile and intravenous anesthetics on pupillary function during general anesthesia in children

DETAILED DESCRIPTION:
The investigator will measure the pupillary function with pupillometry during general anesthesia with volatile or intravenous anesthetics in children.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients undergoing general anesthesia

Exclusion Criteria:

* If injection of any agents that can change pupil size or index
* Any severe side effects, adverse drug reaction

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: From other study results, average NPi for Sevoflurane and propofol were 3.6, 4.2, and standard deviation was 0.1, 0.4 respectively. Using Gpower program, total of 18 patients were required. Considering 20% of drop-out rate, total of 22 patients(18+3.6 patients) were to be recruited.
Sampling Method: Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
NPi | 1hour afer skin incision
  Neurological Pupil index

SECONDARY OUTCOMES:
%CH | 1. Stage of loss of consciousness after induction with bolus propofol 2. Before and after tracheal intubation 3. Skin incision 4. 1hour afer skin incision 5. Just before extubation
  % change of pupil size
CV | 1. Stage of loss of consciousness after induction with bolus propofol 2. Before and after tracheal intubation 3. Skin incision 4. 1hour afer skin incision 5. Just before extubation
  Constriction Velocity
DV | 1. Stage of loss of consciousness after induction with bolus propofol 2. Before and after tracheal intubation 3. Skin incision 4. 1hour afer skin incision 5. Just before extubation
  Dilation Velocity
NPi | 1. Stage of loss of consciousness after induction with bolus propofol 2. Before and after tracheal intubation 3. Skin incision 4. 1hour afer skin incision 5. Just before extubation
  Neurological Pupil index

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No